CLINICAL TRIAL: NCT00779506
Title: A 8-week, Multi-Centre, Open-label, Non-comparative, Phase IV Study of the Efficacy and Safety of Quetiapine Fumarate Extended Release (Seroquel XR) With Daily Dose 400mg-800mg in the Treatment of Acute Schizophrenic Patients
Brief Title: Study of the Efficacy and Safety of Quetiapine Fumarate Extended Release (Seroquel XR)
Acronym: QUENCH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1443L00062
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Results first posted 2011-11-23 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2010-05

CONDITIONS: Schizophrenia
Keywords: Acute schizophrenia; PANSS
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Quetiapine Fumarate XR (Experimental): Seroquel XR 400-800mg
  Interventions: Drug: Quetiapine Fumarate XR

INTERVENTIONS:
Drug: Quetiapine Fumarate XR — oral, once daily, flexible dose
  Other Names: Seroquel XR

SUMMARY:
This is an 8-week, multi-centre, Open-label, non-comparative study to evaluate the efficacy and safety of Quetiapine XR with daily dose 400mg-800mg used as mono-therapy in the treatment of acute schizophrenic patients. The eligible patient will be assigned to study treatment with Quetiapine XR on Day 1.

PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* Documented clinical diagnosis meeting the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) criteria
* PANSS total score of at least 70 at enrolment and at assignment Day 1
* CGI Severity of Illness score of at least 4 (moderately ill) at enrolment and at assignment Day 1 and with worsening of the patient's condition during the 3 weeks

Exclusion Criteria:

* Known intolerance or lack of response to quetiapine fumarate
* Administration of a depot antipsychotic injection within one dosing interval (for the depot) before assignment
* Substance or alcohol dependence at enrolment
* Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 4 weeks prior to enrolment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2008-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: YounHoon Kim, Principal Investigator — Inje University
Locations (7):
- South Korea (7):
  - Research site, Ansan, Gyeonggi-do
  - Research site, Gwangju, Gyeonggi-do
  - Research site, Bugok, Gyeongsangnam-do
  - Research site, Masan, Gyeongsangnam-do
  - Research site, Incheon
  - Research site, Pusan
  - Research site, Seoul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 4 Nov 2008 to 9 July 2009, 96 subjects were enrolled from 9 centers in Korea
Groups:
- Quetiapine XR: This is an 8-week, multi-centre, open-label, non-comparative study to evaluate the efficacy and safety of Quetiapine XR with daily dose 400mg-800mg used as mono-therapy in the treatment of acute schizophrenic patients
Period: Overall Study
Arm/Group | Quetiapine XR
Started | 96
Enrolled | 96
Screen Failed | 2
Assigned | 94
MITT | 89
Treatment Complete | 67
Withdrawal Treatment | 27
Completed | 67
Not Completed | 29
Not completed — Screening Failed | 2
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 11
Not completed — Protocol Violation | 5
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Quetiapine XR
Number analyzed (Participants) | 89
Age Continuous [Mean (Standard Deviation); unit: Years]
  Female | 35.8 (13)
  Male | 42.4 (9.8)
  Total | 39.7 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 52
BMI [Mean (Standard Deviation); unit: kg/m2]
  Female | 23.7 (5.4)
  Male | 23.4 (3.5)
  Total | 23.5 (4.4)
Height [Mean (Standard Deviation); unit: cm]
  Female | 158 (5.9)
  Male | 168.7 (6.6)
  Total | 164.2 (8.2)
Weight [Mean (Standard Deviation); unit: kg]
  Female | 59.1 (13)
  Male | 66.6 (11.4)
  Total | 63.5 (12.6)

OUTCOME MEASURES:

1. Primary Outcome: The Change in Positive and Negative Syndrome Scale(PANSS)Total Score
Description: PANSS, a 30-item scale where each symptom is rated on a severity scale ranging from 1 (absent) - 7 (extreme), total score is 30 - 210.
  Description of the reporting Groups: Evaluate the efficacy of Quetiapine XR with daily dose 400 mg - 800 mg used as mono-therapy in the treatment of acute schizophrenic patients by evaluation of the change from baseline to Day 57 in total score of PANSS using the last observation carried forward (LOCF) method
Time Frame: From baseline to Day 57
Population: The MITT set was used for primary analyses (89) participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quetiapine XR
Number analyzed (Participants) | 89
score on a scale | -26.8 (4.2)

2. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS) Positive Score
Description: To evaluate the change of positive symptoms from baseline to Day 57 in PANSS positive score, a 7-item scale where eash symptom is rated on a severity scale ranging from 1 (absent) - 7 (extreme)
Time Frame: From baseline to Day 57
Population: The MITT set was used for primary analyses (89) participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quetiapine XR
Number analyzed (Participants) | 89
score on a scale | -7.4 (1.2)

3. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS) Negative Score
Description: To evaluate the change of negative symptoms from baseline to Day 57 in PANSS negative score, a 7-item scale where each symptom is rated on a severity scale ranging from 1 (absent) - 7 (extreme)
Time Frame: From baseline to Day 57
Population: The MITT set was used for primary analyses (89) participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quetiapine XR
Number analyzed (Participants) | 89
score on a scale | -6.2 (1.3)

4. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS) General Psychopathology Score
Description: To evaluate the change of general psychopathology symptoms from baseline to Day 57 in PANSS general score, a 16-item scale where each symptom is rated on a severity scale ranging from 1 (absent) to - 7 (extreme)
Time Frame: From baseline to Day 57
Population: The MITT set was used for primary analyses (89) participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quetiapine XR
Number analyzed (Participants) | 89
score on a scale | -13.2 (2.3)

5. Secondary Outcome: Clinical Global Impression (CGI) Score
Description: The Clinical Global Impression - Severity (CGI-S) and - illness (CGI-I) is used in this study. The CGI-S is scored to rate the patient's current clinical state. The CGI-I is scored to rate the patient's change from baseline CGI. Each CGI item is scored on a scale from 1 to 7 (CGI-S: 1 = Normal, not ill, 7= Among the most extremely ill patients/ CGI-I: 1= very much improved, 7= very much worse). CGI-I scores greater than 4 indicate worsening, while scores less than 4 indicate improvement
Time Frame: From baseline to Day 57
Population: The MITT set was used for primary analyses (89) participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quetiapine XR
Number analyzed (Participants) | 89
score on a scale | -1.46 (0.25)

6. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: To treat depressive symptoms in acute schizophrenic patients by evaluation of the change from baseline to day 67 in MADRS total score, a 10-item scale for the evaluation of depressive symptoms. Each MADRS item is rated on a 0-6 scale, higher MADRS scores indicate higher levels of depressive symptoms.
Time Frame: From baseline to Day 57
Population: The MITT set was used for primary analyses (89) participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quetiapine XR
Number analyzed (Participants) | 89
score on a scale | -9.44 (2)

7. Secondary Outcome: Global Assessment of Functioning (GAF) Score
Description: To improve functional capability in acute schizophrenic patients by evaluation of the change from baseline to Day 57 in GAF scale score, a single-item rating scale for evaluating the overall functioning on a continuum from psychologic or psychiatric sickness to health.
Time Frame: From baseline to Day 57
Population: The MITT set was used for primary analyses (89) participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quetiapine XR
Number analyzed (Participants) | 81
score on a scale | 17.9 (2.9)

ADVERSE EVENTS:
Description: Safety population who were taking at least one dose of study treatment were used for the safety analyses (94) participants
Arm/Group | Quetiapine XR
Serious Adverse Events (participants affected / at risk) | 0/94
Other Adverse Events (participants affected / at risk) | 94/94
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine XR (N=94)
Insomnia (Psychiatric disorders) | 22
Anxiety (Psychiatric disorders) | 11
Agitation (Psychiatric disorders) | 5
Constipation (Gastrointestinal disorders) | 24
Dyspepsia (Gastrointestinal disorders) | 9
Toothache (General disorders) | 5
Sedation (Nervous system disorders) | 12
Headache (Nervous system disorders) | 8
Dizziness (Nervous system disorders) | 5
Dysuria (Renal and urinary disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less